CLINICAL TRIAL: NCT02877251
Title: Mexican Multidisciplinary Registry of Patients With Venous Thromboembolic Disease
Acronym: REMMITE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Registro Mexicano Multidisciplinario De Pacientes Con Enfermedad Tromboembolica Venosa (Other)
Collaborators: Webmedica (Unknown)
Responsible Party: Sponsor
Other Study IDs: REMMITE
Record Dates: First submitted 2016-08-12; First posted 2016-08-24 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism
Keywords: Venous Thromboembolism; Venous Thrombosis; Pulmonary Thromboembolism; National Registry; Mexico; Major Adverse Cardiovascular Events
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Deep venous thrombosis: To identify clinical characteristics, treatment trends, in-hospital and 3, 6, and 12 months follow-up outcome through major adverse cardiovascular events (MACE) of patients diagnosed with deep venous thrombosis
- Deep venous thrombosis and Pulmonary embolism: To identify clinical characteristics, treatment trends, in-hospital and 3, 6, and 12 months follow-up outcome through major adverse cardiovascular events (MACE) of patients diagnosed with deep venous thrombosis and pulmonary embolism
- Pulmonary embolism: To identify clinical characteristics, treatment trends, in-hospital and 3, 6, and 12 months follow-up outcome through major adverse cardiovascular events (MACE) of patients diagnosed with pulmonary embolism

SUMMARY:
REMMITE, a retrospective and prospective registry with one-year follow-up, will provide valuable insights into the clinical diagnosis, management, treatment trends as well as related outcomes of three cohorts: DVT, DVT-PE, PE patients throughout many regions of Mexico and through different health care systems.

DETAILED DESCRIPTION:
Introduction Venous thromboembolism disease, (VTE) comprises deep venous thrombosis (DVT) and pulmonary embolism (PE). In United States, incidence has remained relatively constant. In Mexico, annual incidence is unknown. In spite of technological and risk stratification advances, it is still the third cause of cardiovascular and pulmonary disease. Presentation of PE is quite heterogeneous. As a complex disease with highly variable presentations in different clinical settings, DVT-PE can be confronted and managed by cardiologists, pneumologists, intensive care, internal medicine, emergency, orthopedics and surgery physicians. Thus, initial clinical approach and results can vary depending on attending physicians, experience and hospital infrastructure.

The mainstay of VTE treatment is anticoagulation, either systemic or oral. PE management, however, varies widely, depending on patient presentation but substantially on hemodynamic consequences based of right ventricle (RV) dysfunction. A careful clinical history and physical examination, integrated to electrocardiographic, laboratory and appropriate imaging findings could help to risk stratification in order to proceed to a treatment. Though some patients present with clear hemodynamic compromise, others may have an incidentally diagnosis while a test is performed for a different reason. Scoring systems can identify patients at different levels of risk. Registries may help to get key findings to quantify clinical characteristics, electrocardiographic, laboratory and modality imaging as well as treatment trends and clinical outcomes in the real world.

Results of the REMMITE, a retrospective and prospective registry with one-year follow-up, will provide valuable insights into the clinical diagnosis, management, treatment trends as well as related outcomes. The REMMITE has the potential to dictate guidelines and recommendations based on identified deficits and good practices among participating centers.

REMMITE design Primary objective: to identify clinical characteristics, treatment trends, in-hospital and 12 months follow-up outcome through major adverse cardiovascular events (MACE) of patients diagnosed either with DVT, DVT-PE, or PE.

Variables to be included In all patients: a) demographic data, b) date of onset of symptoms, c) past medical history, d) physical examination e) electrocardiographic, f) laboratory and g) imaging findings, h) treatment in acute phase, i) in-hospital and follow - up outcome, j) treatment during follow-up, k) MACE.

Retrospective cases enrollment Patients with a history of DVT, DVT-PE, PE in the last year will be enrolled. In all patients: a) demographic data, b) date of onset of symptoms, c) past medical history, d) physical examination e) electrocardiographic, f) laboratory and g) imaging findings, h) treatment in acute phase, i) in-hospital and follow - up outcome, j) treatment during follow-up, in patients under oral anticoagulation with vitamin K antagonists International Normalized Ratio (INR) will be recorded; k) percentage of patients with non-vitamin K antagonist (NOAC´s) during following) l) MACE.

Prospective cases enrollment Patients with an acute episode of DVT, DVT-PE, PE will be enrolled. In all patients: a) demographic data, b) date of onset of symptoms, c) past medical history, d) physical examination e) electrocardiographic, f) laboratory and g) imaging findings, h) treatment in acute phase, i) in-hospital and follow - up outcome, j) treatment during follow-up,( in patients under oral anticoagulation with vitamin K antagonists INR will be recorded;) k) patients receiving (NOAC´s) drugs at discharge, l) percentage of patients with NOAC´s during following, m) MACE.

Sites Centers with investigators with expertise in diagnosis, stratification and treatment of patients with DVT, DVT-PE, PE will be involved. Also, Centers without expertise, but with facilities to diagnosis and treatment and real interest in enrolling will be included, as long as they accomplish with protocol requirements.

Quality Criteria Following criteria will be used to guarantee quality data: a) electronic, simple and accessible data collection, back-upped by clinical file, b) participate in a assay filling to be familiar with electronic data collection, c) standardized definitions, data and reports; d) meetings among principal investigators and steering committee at least once a year; e) ethics procedures review; f) rigorous center selection based on investigators expertise and/or facilities resources); g) consecutive patients enrollment to obtain representative sample; h) random centers audit; i) centralized data and statistical analysis; j) report all data and consistent conclusion; and k) transparency of funds for any publication. Also, a way to qualify quality of this registry will be measured by the number of publications and presentations in national and international meetings.

Data collection Electronic database will have specific variables such as: date of onset symptoms, medical history, personal history, physical examination, electrocardiographic, chest x-Ray, echocardiogram, V/Q lung scan, magnetic resonance imaging, chest computed tomography, pulmonary angiography, right heart catheterization, venous ultrasound, biomarkers, treatment either pharmacologic or percutaneous, and MACE.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years;
* clinical diagnosis of DVT, DVT-PE, PE.

Exclusion Criteria:

* chronic DVT;
* chronic PE;
* refusal to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DVT, DVT-PE, PE patients throughout many regions of Mexico and through different health care systems.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  to identify clinical characteristics, treatment trends, in-hospital and 12 months follow-up outcome through major adverse cardiovascular events (MACE) of patients diagnosed either with DVT, DVT-PE, or PE.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gutierrez-Fajardo, MD, Principal Investigator